CLINICAL TRIAL: NCT06386471
Title: Personalized Gastrointestinal Motility Responses to Dietary Fiber and Gut Microbial Metabolites
Brief Title: Personalized GI Motility Responses to Diet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24093
Record Dates: First submitted 2024-03-04; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Nutritional and Metabolic Diseases; Gastrointestinal Dysfunction; Cardiovascular Diseases; Dysbiosis
Keywords: dietary fiber; gastrointestinal motility; cardiometabolic; microbiome
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Cardiovascular Diseases; Dysbiosis

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, crossover
Masking Description: Appearance, flavor, and texture of whole grain vs refined bread could not be masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole grain rye bread (Experimental): 4.3 ounces of whole grain rye bread, consumed after an overnight fast (12+ hours)
  Interventions: Other: Whole grain rye bread
- Refined grain rye bread (Placebo Comparator): 4.3 ounces of white rye bread, consumed after an overnight fast (12+ hours)
  Interventions: Other: Refined grain rye bread

INTERVENTIONS:
Other: Whole grain rye bread — Single consumption of 4.3 oz of whole grain rye bread
  Arms: Whole grain rye bread
Other: Refined grain rye bread — Single consumption of 4.3 oz of refined grain rye bread
  Arms: Refined grain rye bread

SUMMARY:
The goal of this randomized, crossover, clinical trial is to link: 1) gastrointestinal motility patterns induced by acute consumption of whole and refined grains, 2) enteric microbial production of bioactive metabolites, and 3) circulating postprandial appearance of metabolites important to cardiometabolic health including glucose, triglycerides, and cholesterol.

Participants will be asked to consume a Smartpill monitoring device that records metrics of gastrointestinal motility in response to whole or refined grains, monitor cardiometabolic metabolties over an 8 hour postprandial window, and provide a fecal sample for microbiome-related analyses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women

Exclusion Criteria:

Physician-Diagnosed:

* Diabetes Mellitus
* Nutrient-malabsorption disorders
* Intestinal Bowel Syndrome (IBS)
* Intestinal Bowel Disease (IBD)
* Bleeding-related disorders
* Grain allergy
* Psychological Disorders
* Stenosis
* Dysphasia

History of:

* Bariatric Surgery
* Gallbladder removal
* Eating disorders
* Antibiotic administration (within the past three months)
* Hormone therapy

Currently:

* Using statins
* Pregnant, lactating, or postmenopausal
* Taking oral hypoglycemic agents or insulin
* Ingesting prescription fiber
* Using cholesterol and bile acid absorption inhibitors
* Ingesting nutrition supplements, not including a daily multivitamin (i.e. herbs, tinctures, and extracts) •Using recreational drugs or alcohol (within the past week)
* Taking anti-histamines
* Taking proton pump inhibitors
* Taking antacids

Ages: 21 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-06-12 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Pressure (mmHg) | From consumption of bread and Smartpill to deification (single meal consumption, GI motility times vary based on participant, but could be estimated from around 16 hours to 5 days)
  Pressure of gastrointestinal contractions as captured by the Medtronic Smartpill capsule temperature, transit time)
Luminal pH (pH units) | From consumption of bread and Smartpill to deification (single meal consumption, GI motility times vary based on participant, but could be estimated from around 16 hours to 5 days)
  pH of gastrointestinal contents as captured by the Medtronic Smartpill capsule
Temperature (degrees celcius) | From consumption of bread and Smartpill to deification (single meal consumption, GI motility times vary based on participant, but could be estimated from around 16 hours to 5 days)
  Temperature in the intestinal lumen as captured by the Medtronic Smartpill capsule
Gastrointestinal Transit Time (hours:minutes) | From consumption of bread and Smartpill to deification (single meal consumption, GI motility times vary based on participant, but could be estimated from around 16 hours to 5 days)
  Duration of gastrointestinal transit as captured by the Medtronic Smartpill capsule
Blood Glucose | Baseline to 8 hours post bread and Smartpill consumption (baseline, 0.5 hours, 1 hour, 1.5 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, and 8 hours)
  Concentration of glucose in whole blood from finger prick as measured by the Konsung Portable Dry Biochemical Analyzer
Triglycerides | Baseline to 8 hours post bread and Smartpill consumption (baseline, 0.5 hours, 1 hour, 1.5 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, and 8 hours)
  Concentration of triglycerides in whole blood from finger prick as measured by the Konsung Portable Dry Biochemical Analyzer
Total Cholesterol | Baseline to 8 hours post bread and Smartpill consumption (baseline, 0.5 hours, 1 hour, 1.5 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, and 8 hours)
  Concentration of total cholesterol in whole blood from finger prick as measured by the Konsung Portable Dry Biochemical Analyzer
HDL cholesterol | Baseline to 8 hours post bread and Smartpill consumption (baseline, 0.5 hours, 1 hour, 1.5 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, and 8 hours)
  Concentration of HDL cholesterol in whole blood from finger prick as measured by the Konsung Portable Dry Biochemical Analyzer
LDL cholesterol | Baseline to 8 hours post bread and Smartpill consumption (baseline, 0.5 hours, 1 hour, 1.5 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, and 8 hours)
  Concentration of LDL choelsterol in whole blood from finger prick as measured by the Konsung Portable Dry Biochemical Analyzer
Lipopolysaccharide Binding Protein | Baseline to 8 hours post bread and Smartpill consumption (baseline, 0.5 hours, 1 hour, 1.5 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, and 8 hours)
  Concentration of LBP in whole blood from finger prick as measured by ELISA

SECONDARY OUTCOMES:
Microbiome | Fecal sample following ingestion of the Smartpill and test meal (approximately 24 hours into the study arm)
  Shotgun metagenomic sequencing of fecal samples, including metrics of diversity (ex: shannon index), taxonomic abundances (relative abundance, %), functional gene abundances (relative abundance, %), etc
Metabolomics | Fecal sample following ingestion of the Smartpill and test meal (approximately 24 hours into the study arm)
  Untargeted metabolomics of fecal samples via LC-MS, including metrics of pathway analysis (pathway score), single metabolite relative concentration (relative intensity), etc

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States